CLINICAL TRIAL: NCT02226627
Title: Latin American Survey of Nutrition and Health / Estudio Latinoamericano de Nutrición y Salud
Status: Completed | Type: Observational
Sponsor: Mauro Fisberg (Other)
Collaborators: International Life Sciences Institute, Argentina (Unknown); Pontificia Universidad Catolica de Chile (Other); Pontificia Universidad Javeriana (Other); Universidad de Costa Rica (Other); Universidad San Francisco de Quito (Other); Instituto de Investigacion Nutricional, Peru (Other); Universidad Central de Venezuela (Other)
Responsible Party: Sponsor-Investigator, Mauro Fisberg, MD, PhD, Hospital Infantil Sabará
Organization: Hospital Infantil Sabará (Other)
Other Study IDs: ELANS-2014
Record Dates: First submitted 2014-08-22; First posted 2014-08-27 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Dietary Habits; Physical Activity; Overweight and Obesity
MeSH Terms: conditions — Feeding Behavior; Motor Activity; Overweight; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to make a proper scientific assessment on the dietary intake and physical activity levels of a representative sample of the urban population of 8 Latin American countries (Argentina, Brazil, Chile, Colombia, Costa Rica, Ecuador, Perú and Venezuela). The study was based on complex, multistage sample design, stratified by conglomerates, being all regions of each country represented, and random selection of main cities within each region according to probability proportional to size method. Sample will be stratified by gender, age (15 to 65 years old), and socioeconomic level. Socioeconomic levels will be balanced and divided in three strata (high, medium and low) based on national indexes used in each country. All the study sites are university-based and will adhere to a common study protocol for training, implementation of fieldwork, data collection and management, and quality control procedures to be performed simultaneously. All participants will be required to provide a written informed consent. A pilot study at small scale will be performed in each country in order to test procedures and tools involved in ELANS. Anthropometric variables, including body weight, height, waist, hip and neck circumferences will be measured according to a standardized protocol. Nutritional intake evaluation will be performed using two 24-hour dietary recalls, with 'multiple pass' procedure and a food frequency questionnaire. Nutritional data will be entered in Nutrition Data System for Research (NDS-R, Minnesota University) after a harmonization process between local foods and NDSR database. Physical activity and energy expenditure will be assessed by IPAQ-long version questionnaire and 7-day accelerometry.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* 15 to 65 years old

Exclusion Criteria:

* Adolescents without assent and parent´s or legal guardian´s permission will be excluded
* Any adolescent or adult with mental and/or physical disability will be excluded.
* Any adolescent or adult with a chronic or acute illness that may affect normal eating behavior or energy expenditure will be excluded.
* Pregnant and nursing women of a child younger than 6 months will be excluded.
* Any adolescent or adult who is not able to read will be excluded.
* Any adolescent or adult who is not present at or refuses to accept the second visit will be excluded.
* Any adolescent or adult living in any residential settings different from a household (hospitals, regiments, homes, such as old-age homes, etc.) and mobile homes or trailers are excluded.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The sample will include subjects of both sexes, between 15 and 65 years old, considering four age ranges (as see below), that belong to high, middle or low socioeconomic levels (SEL), living in private households in the major cities and other relevant cities in terms of population weight, according to the regions of each of the countries selected for the study.
Sampling Method: Probability Sample
Enrollment: 9000 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
overweight/obesity | baseline
  overweight/obesity will be assessed via anthropometric evaluation
energy intake | 2 food records will be applied with 7 days apart
  Nutritional intake will be performed using two 24-hour dietary recalls, with 'multiple pass' procedure
energy expenditure | 1 week
  accelerometer measurement during 1 week

SECONDARY OUTCOMES:
snack intake | 2 food records will be applied with 7 days apart
  snack intake will be evaluated using two 24-hour dietary recalls, with 'multiple pass' procedure
beverage intake | after 7 days
  Beverage intake will be evaluated using a food frequency questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Fisberg, MD PhD, Principal Investigator — Instituto Pensi- Fundação Jose Luiz Setubal - Hospital Infantil Sabara
Locations (8):
- International Life Science Institute (ILSI), Buenos Aires, Buenos Aires, Argentina
- Instituto Pensi- Fundação Jose Luiz Setubal - Hospital Infantil Sabara, São Paulo, São Paulo, Brazil
- Departamento de Nutrición, Diabetes y Metabolismo, Centro de Nutrición Molecular y Enfermedades Crónicas - Pontificia Universidad Católica, Santiago, Chile
- Departamento de Nutrición y Bioquímica - Pontificia Universidad Javeriana, Bogotá, Colombia
- Departamento de Bioquímica - Escuela de Medicina - Universidad de Costa Rica, San José, Costa Rica
- Universidad San Francisco de Quito, Quito, Ecuador
- Instituto de Investigación Nutricional, Lima, Peru
- Centro de Estudios del Desarrollo - Universidade Central da Venezuela (CENDES-UCV)/Fundación Bengoa, Caracas, Venezuela

REFERENCES:
- [Derived] de Victo ER, Gomez G, Fisberg M, Kovalskys I, Ferrero-Hernandez P, Farias-Valenzuela C, Figueiredo TKF, Ferrari G. Joint associations of accelerometer-measured physical activity and sedentary time with body mass index: Cross-sectional evidence from the Latin American Study of Nutrition and Health. Obes Res Clin Pract. 2025 Jul-Aug;19(4):297-302. doi: 10.1016/j.orcp.2025.08.004. Epub 2025 Aug 14. PMID 40813228
- [Derived] Kloss RF, Lorca JC, Rivera AR, Saldana BF, de Victo ER, Ferrari G. Perceived neighborhood built environment and physical activity in urban population in Chile. BMC Public Health. 2025 Mar 11;25(1):969. doi: 10.1186/s12889-025-22138-z. PMID 40069644
- [Derived] de Victo ER, Fisberg M, Sole D, Kovalskys I, Gomez G, Rigotti A, Cortes LY, Yepez-Garcia MC, Pareja R, Herrera-Cuenca M, Drenowatz C, Christofaro D, Araujo T, Silva D, Ferrari G. Joint Association between Sedentary Time and Moderate-to-Vigorous Physical Activity with Obesity Risk in Adults from Latin America. Int J Environ Res Public Health. 2023 Apr 18;20(8):5562. doi: 10.3390/ijerph20085562. PMID 37107844
- [Derived] de Victo ER, Kovalskys I, Fisberg M, Gomez G, Rigotti A, Cortes LY, Garcia MY, Pareja RG, Herrera-Cuenca M, Sole D, Drenowatz C, Marques A, Ferrari G. Are the different cut-off points for sitting time associated with excess weight in adults? A population based study in Latin America. BMC Public Health. 2023 Jan 16;23(1):110. doi: 10.1186/s12889-023-15029-8. PMID 36647028
- [Derived] Villar M, Garcia MCY, Ocampo MB, Gomez G. Intake and food sources of sodium in the population residing in urban areas of Ecuador: results from ELANS study. Glob Health Action. 2023 Dec 31;16(1):2156110. doi: 10.1080/16549716.2022.2156110. PMID 36601889
- [Derived] Ferrari G, Drenowatz C, Kovalskys I, Gomez G, Rigotti A, Cortes LY, Garcia MY, Pareja RG, Herrera-Cuenca M, Del'Arco AP, Peralta M, Marques A, Leme ACB, Sadarangani KP, Guzman-Habinger J, Chaves JL, Fisberg M. Walking and cycling, as active transportation, and obesity factors in adolescents from eight countries. BMC Pediatr. 2022 Aug 30;22(1):510. doi: 10.1186/s12887-022-03577-8. PMID 36042429
- [Derived] Ferrari G, Farias-Valenzuela C, Guzman-Habinger J, Drenowatz C, Marques A, Kovalskys I, Gomez G, Rigotti A, Cortes LY, Yepez Garcia MC, Pareja RG, Herrera-Cuenca M, Marconcin P, Chavez JL, Fisberg M. Relationship between socio-demographic correlates and human development index with physical activity and sedentary time in a cross-sectional multicenter study. BMC Public Health. 2022 Apr 6;22(1):669. doi: 10.1186/s12889-022-13117-9. PMID 35387627
- [Derived] Yepez Garcia MC, Herrera-Cuenca M, Ferrari G, Sanabria LYC, Hernandez P, Almeida RY, Villar Caceres M, Gomez G, Pareja R, Rigotti A, Kovalskys I, Fisberg M. Energy Imbalance Gap, Anthropometric Measures, Lifestyle, and Sociodemographic Correlates in Latin American Adults-Results from the ELANS Study. Int J Environ Res Public Health. 2022 Jan 20;19(3):1129. doi: 10.3390/ijerph19031129. PMID 35162152
- [Derived] Ferrari G, Alberico C, Drenowatz C, Kovalskys I, Gomez G, Rigotti A, Cortes LY, Garcia MY, Liria-Dominguez MR, Herrera-Cuenca M, Peralta M, Marques A, Marconcin P, Cristi-Montero C, Leme ACB, Zimberg IZ, Farias-Valenzuela C, Fisberg M, Rollo S. Prevalence and sociodemographic correlates of meeting the Canadian 24-hour movement guidelines among latin american adults: a multi-national cross-sectional study. BMC Public Health. 2022 Feb 3;22(1):217. doi: 10.1186/s12889-022-12613-2. PMID 35109819
- [Derived] Ferrari G, Werneck AO, Silva DR, Kovalskys I, Gomez G, Rigotti A, Cortes LY, Garcia MCY, Liria-Dominguez MR, Herrera-Cuenca M, Pratt M, Marques A, Van Dyck D, Leme ACB, Fisberg M. Perceived Urban Environment Attributes and Device-Measured Physical Activity in Latin America: An 8-Nation Study. Am J Prev Med. 2022 Apr;62(4):635-645. doi: 10.1016/j.amepre.2021.09.006. Epub 2021 Nov 19. PMID 34810040
- [Derived] Barreno M, Sisa I, Yepez Garcia MC, Shen H, Villar M, Kovalskys I, Fisberg M, Gomez G, Rigotti A, Cortes LY, Pareja RG, Herrera-Cuenca M, Guajardo V; ELANS Study Group. Association between built environment and physical activity in Latin American countries: a multicentre cross-sectional study. BMJ Open. 2021 Nov 3;11(11):e046271. doi: 10.1136/bmjopen-2020-046271. PMID 34732475
- [Derived] Ferrari G, Guzman-Habinger J, Chavez JL, Werneck AO, Silva DR, Kovalskys I, Gomez G, Rigotti A, Cortes LY, Yepez Garcia MC, Pareja RG, Herrera-Cuenca M, Drenowatz C, Cristi-Montero C, Marques A, Peralta M, Leme ACB, Fisberg M. Sociodemographic inequities and active transportation in adults from Latin America: an eight-country observational study. Int J Equity Health. 2021 Aug 26;20(1):190. doi: 10.1186/s12939-021-01524-0. PMID 34446008
- [Derived] Del'Arco APWT, Previdelli AN, Ferrari G, Fisberg M. Food intake, physical activity and body composition of adolescents and young adults: data from Brazilian Study of Nutrition and Health. BMC Public Health. 2021 Jun 12;21(1):1123. doi: 10.1186/s12889-021-11171-3. PMID 34118909
- [Derived] Ferrari G, Marques A, Barreira TV, Kovalskys I, Gomez G, Rigotti A, Cortes LY, Garcia MCY, Pareja RG, Herrera-Cuenca M, Guajardo V, Leme ACB, Guzman Habinger J, Valdivia-Moral P, Suarez-Reyes M, Ihle A, Gouveia ER, Fisberg M, On Behalf Of The Elans Study Group. Accelerometer-Measured Daily Step Counts and Adiposity Indicators among Latin American Adults: A Multi-Country Study. Int J Environ Res Public Health. 2021 Apr 27;18(9):4641. doi: 10.3390/ijerph18094641. PMID 33925513
- [Derived] Ferrari G, Werneck AO, Silva DR, Kovalskys I, Gomez G, Rigotti A, Cortes LY, Garcia MY, Liria M, Herrera-Cuenca M, Zimberg IZ, Guajardo V, Pratt M, Cristi-Montero C, Marques A, Peralta M, Bolados CC, Leme ACB, Rollo S, Fisberg M; ELANS Study Group. Agreement Between Self-Reported and Device-Based Sedentary Time among Eight Countries: Findings from the ELANS. Prev Sci. 2021 Nov;22(8):1036-1047. doi: 10.1007/s11121-021-01206-x. Epub 2021 Jan 27. PMID 33502675
- [Derived] Ferrari G, Werneck AO, da Silva DR, Kovalskys I, Gomez G, Rigotti A, Sanabria LYC, Garcia MY, Pareja RG, Herrera-Cuenca M, Zimberg IZ, Guajardo V, Pratt M, Cristi-Montero C, Rodriguez-Rodriguez F, Marques A, Cerin E, Van Dyck D, Pires C, Fisberg M; ELANS Study Group. Is the perceived neighborhood built environment associated with domain-specific physical activity in Latin American adults? An eight-country observational study. Int J Behav Nutr Phys Act. 2020 Oct 1;17(1):125. doi: 10.1186/s12966-020-01030-6. PMID 33004078
- [Derived] Ferrari GLM, Oliveira Werneck A, Rodrigues da Silva D, Kovalskys I, Gomez G, Rigotti A, Yadira Cortes Sanabria L, Garcia MCY, Pareja RG, Herrera-Cuenca M, Zalcman Zimberg I, Guajardo V, Pratt M, Cofre Bolados C, Fuentes Kloss R, Rollo S, Fisberg M. Socio-Demographic Correlates of Total and Domain-Specific Sedentary Behavior in Latin America: A Population-Based Study. Int J Environ Res Public Health. 2020 Aug 3;17(15):5587. doi: 10.3390/ijerph17155587. PMID 32756330
- [Derived] Ferrari GLM, Kovalskys I, Fisberg M, Gomez G, Rigotti A, Sanabria LYC, Garcia MCY, Torres RGP, Herrera-Cuenca M, Zimberg IZ, Guajardo V, Pratt M, Previdelli AN, Scholes S, Celis-Morales CA, Sole D; ELANS Study Group. Anthropometry, dietary intake, physical activity and sitting time patterns in adolescents aged 15-17 years: an international comparison in eight Latin American countries. BMC Pediatr. 2020 Jan 21;20(1):24. doi: 10.1186/s12887-020-1920-x. PMID 31964386
- [Derived] Luis de Moraes Ferrari G, Kovalskys I, Fisberg M, Gomez G, Rigotti A, Sanabria LYC, Garcia MCY, Torres RGP, Herrera-Cuenca M, Zimberg IZ, Guajardo V, Pratt M, King AC, Sole D; ELANS Study Group. Original research Socio-demographic patterning of self-reported physical activity and sitting time in Latin American countries: findings from ELANS. BMC Public Health. 2019 Dec 23;19(1):1723. doi: 10.1186/s12889-019-8048-7. PMID 31870408
- [Derived] Luis de Moraes Ferrari G, Kovalskys I, Fisberg M, Gomez G, Rigotti A, Sanabria LYC, Garcia MCY, Torres RGP, Herrera-Cuenca M, Zimberg IZ, Guajardo V, Pratt M, Pires C, Sole D; ELANS Study Group. Association of moderate-to-vigorous physical activity with neck circumference in eight Latin American countries. BMC Public Health. 2019 Jun 24;19(1):809. doi: 10.1186/s12889-019-7153-y. PMID 31234866
- [Derived] Kovalskys I, Fisberg M, Gomez G, Pareja RG, Yepez Garcia MC, Cortes Sanabria LY, Herrera-Cuenca M, Rigotti A, Guajardo V, Zalcman Zimberg I, Nogueira Previdelli A, Moreno LA, Koletzko B; ELANS Study Group. Energy intake and food sources of eight Latin American countries: results from the Latin American Study of Nutrition and Health (ELANS). Public Health Nutr. 2018 Oct;21(14):2535-2547. doi: 10.1017/S1368980018001222. Epub 2018 May 31. PMID 29848396
- [Derived] Fisberg M, Kovalskys I, Gomez G, Rigotti A, Cortes LY, Herrera-Cuenca M, Yepez MC, Pareja RG, Guajardo V, Zimberg IZ, Chiavegatto Filho ADP, Pratt M, Koletzko B, Tucker KL; ELANS Study Group. Latin American Study of Nutrition and Health (ELANS): rationale and study design. BMC Public Health. 2016 Jan 30;16:93. doi: 10.1186/s12889-016-2765-y. PMID 26829928